CLINICAL TRIAL: NCT02460679
Title: A Phase 2A Safety and Biomarker Study of EPI-589 in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Safety and Biomarker Study of EPI-589 in Participants With Amyotrophic Lateral Sclerosis (ALS)
Acronym: EPI-589
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI589-15-001
Record Dates: First submitted 2015-05-21; First posted 2015-06-02 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EPI-589 (Experimental): Participants will receive EPI-589 500 milligrams (mg) (2 tablets of 250 mg each) twice daily (BID) for 3 months, unless discontinued for safety or tolerability issues.
  Interventions: Drug: EPI-589

INTERVENTIONS:
Drug: EPI-589 — An immediate release film-coated table at a 250 mg dosage strength will be administered per dose and schedule specified in arm.
  Other Names: (R)-troloxamide quinone

SUMMARY:
This is an open label study with 30-day run in phase to establish baseline parameters, 90-day treatment phase, and a 90-day withdrawal phase to determine long-term effects, duration of treatment response, and potential effects of EPI-589 therapy on known trajectory.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable, laboratory supported probable, or definite ALS by E1 Escorial Criteria
* Forced vital capacity (FVC) ≥ 70% of predicted
* Weakness onset within 3 years
* Agreement to use contraception if within reproductive years
* Willingness and ability to comply with study procedures
* Stable regimen of dietary supplements and /or riluzole for at least 30 days prior to enrollment
* Abstention from use of other investigative or non-approved drugs
* Participants must be able to swallow 0.375 * 0.700 inch tablets

Exclusion Criteria:

* Allergy to EPI-589
* Use of ventilation
* Participation in other intervention studies
* Diagnosis of any other neurologic disease
* Malignancy within the past 2 years
* History of stroke
* History of brain surgery
* Hepatic insufficiency with liver function tests (LFTs) greater than 3 times upper limit of normal (ULN)
* Renal insufficiency requiring dialysis
* End stage cardiac failure
* Participation in a trial of a device, drug, or other therapy for ALS within 3 months of screening or during the trial

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Klein, MD, FACS, Study Director — PTC Therapeutics
Locations (3):
- United States (3):
  - Cedar's Sinai, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Providence Brain and Spine Institute ALS Center, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- EPI-589: Participants received EPI-589 500 milligrams (mg) (2 tablets of 250 mg each) twice daily (BID) for 3 months, unless discontinued for safety or tolerability issues.
Period: Overall Study
Arm/Group | EPI-589
Started | 19
Received at Least 1 Dose of Study Drug | 19
Completed | 14
Not Completed | 5
Not completed — Investigator Decision | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Efficacy intent-to-treat (EITT) population or safety population included any participant who received at least 1 dose of EPI-589.
Groups:
- EPI-589: Participants received EPI-589 500 mg (2 tablets of 250 mg each) BID for 3 months, unless discontinued for safety or tolerability issues.
Arm/Group | EPI-589
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) Score [Mean (Standard Deviation); unit: units on a scale] — ALSFRS-R is a quickly administered (5 minutes) ordinal rating scale that assesses participant's capability and independence in 12 functional activities. All 12 activities, 6 bulbar-respiratory functions, 3 upper extremity functions (writing, cutting food, and dressing), 2 lower-extremity functions (walking and climbing), and 1 other function (turning in bed), are relevant in amyotrophic lateral sclerosis (ALS). Each activity was recorded to the closest approximation from a list of 5 choices, scored 0-4, with the total score ranging from 48 (normal function) to 0 (unable to attempt the task).
  units on a scale | 37.4 (6.19)
Vital Capacity [Mean (Standard Deviation); unit: percentage of capacity] — Vital capacity is the maximum amount of air a participant can expel from the lungs after a maximum inhalation.
  percentage of capacity | 97.7 (18.14)
Maximum Inspiratory Pressure (MIP) [Mean (Standard Deviation); unit: centimetres of water at (cm H2O)] — MIP is a measure of the strength of inspiratory muscles, primarily the diaphragm, and allows for the assessment of ventilatory failure, restrictive lung disease, and respiratory muscle strength.
  centimetres of water at (cm H2O) | 68.2 (34.53)
Respiratory Rate [Mean (Standard Deviation); unit: breaths/minute] — Respiratory rate is the rate at which breathing occurs. Population: 'Number analyzed' signifies participants evaluable for specified categories.
  breaths/minute
    Sitting | 15.1 (3.32)
    After 5 minutes supine: number analyzed (Participants) | 13
    After 5 minutes supine | 14.7 (3.71)
    After 10 minutes supine: number analyzed (Participants) | 15
    After 10 minutes supine | 14.7 (3.28)
Heart Rate [Mean (Standard Deviation); unit: beats/minute] — The heart rate measures the number of times the heart beats per minute. Population: 'Number analyzed' signifies participants evaluable for specified categories.
  beats/minute
    Sitting | 68.9 (10.99)
    After 5 minutes supine: number analyzed (Participants) | 13
    After 5 minutes supine | 63.8 (13.46)
    After 10 minutes supine: number analyzed (Participants) | 15
    After 10 minutes supine | 65.3 (12.30)
Oxygen Saturation (SpO2) [Mean (Standard Deviation); unit: percentage of hemoglobin] — SpO2, also known as oxygen saturation, is a measure of the amount of oxygen-carrying hemoglobin in the blood relative to the amount of hemoglobin not carrying oxygen. Population: 'Number analyzed' signifies participants evaluable for specified categories.
  percentage of hemoglobin
    Sitting | 96.9 (1.65)
    After 5 minutes supine: number analyzed (Participants) | 13
    After 5 minutes supine | 95.4 (2.79)
    After 10 minutes supine: number analyzed (Participants) | 15
    After 10 minutes supine | 95.1 (2.70)
End-Tidal Carbon Dioxide (ETCO2) [Mean (Standard Deviation); unit: percentage of CO2] — ETCO2 is the amount of CO2 in exhaled air, which assesses ventilation. Population: 'Number analyzed' signifies participants evaluable for specified categories.
  percentage of CO2
    Sitting | 24.833 (16.8444)
    After 5 minutes supine: number analyzed (Participants) | 13
    After 5 minutes supine | 30.964 (15.9007)
    After 10 minutes supine: number analyzed (Participants) | 15
    After 10 minutes supine | 31.186 (14.5895)
Average Solid Swallowing Time [Mean (Standard Deviation); unit: seconds] | 12.46 (5.465)
Average Water Swallowing Time [Mean (Standard Deviation); unit: seconds] | 4.68 (3.698)
Muscle Function, as Assessed by Handheld Dynamometry Parameters [Mean (Standard Deviation); unit: kilograms] — Handheld dynamometry parameters included grip strength, shoulder flexion, knee extension, hip flexion, elbow flexion, elbow extension, and ankle dorsi flexion. Population: 'Number analyzed' signifies participants evaluable for specified categories.
  kilograms
    Grip - Left: number analyzed (Participants) | 17
    Grip - Left | 26.41 (20.630)
    Grip - Right: number analyzed (Participants) | 18
    Grip - Right | 26.86 (18.667)
    Shoulder Flexion - Left: number analyzed (Participants) | 17
    Shoulder Flexion - Left | 13.94 (8.218)
    Shoulder Flexion - Right: number analyzed (Participants) | 17
    Shoulder Flexion - Right | 14.42 (9.850)
    Knee Extension - Left | 22.11 (12.796)
    Knee Extension - Right | 22.13 (13.224)
    Knee Flexion - Left | 17.32 (11.832)
    Knee Flexion - Right | 18.02 (12.987)
    Hip Flexion - Left | 20.13 (16.229)
    Hip Flexion - Right | 20.82 (12.738)
    Elbow Flexion - Left: number analyzed (Participants) | 17
    Elbow Flexion - Left | 17.16 (9.074)
    Elbow Flexion - Right: number analyzed (Participants) | 17
    Elbow Flexion - Right | 16.52 (10.508)
    Elbow Extension - Left: number analyzed (Participants) | 17
    Elbow Extension - Left | 17.51 (10.514)
    Elbow Extension - Right: number analyzed (Participants) | 18
    Elbow Extension - Right | 15.36 (10.482)
    Ankle Dorsi Flexion - Left: number analyzed (Participants) | 18
    Ankle Dorsi Flexion - Left | 16.47 (12.188)
    Ankle Dorsi Flexion - Right: number analyzed (Participants) | 18
    Ankle Dorsi Flexion - Right | 13.04 (10.898)
Number of Words Participant Read [Mean (Standard Deviation); unit: Words] | 100.3 (0.45)
Time Spent in Reading [Mean (Standard Deviation); unit: seconds] | 48.5 (23.51)
Number of Words Per Minute Read [Mean (Standard Deviation); unit: words/minute] | 143.529 (45.4527)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-Related Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline (Day 0) to Month 6
Population: Safety population included any participant who received at least 1 dose of EPI-589.
Measure: Count of Participants; unit: Participants
Arm/Group | EPI-589
Number analyzed (Participants) | 19
Participants | 0

2. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 12 Hours (AUC0-12)
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose at Month 1 and 3
Population: EITT population or safety population included any participant who received at least 1 dose of EPI-589. Here, 'Number analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Standard Error); unit: hours*nanograms/milliliter
Arm/Group | EPI-589
Number analyzed (Participants) | 19
hours*nanograms/milliliter
  Month 1: number analyzed (Participants) | 10
  Month 1 | 7762.7 (721.1)
  Month 3: number analyzed (Participants) | 9
  Month 3 | 6878.8 (401.1)

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose (0 hour), 0.5, 1, 2, 4, 6, 8, and 12 hours post-dose at Month 1 and 3
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | EPI-589
Number analyzed (Participants) | 19
ng/mL
  Month 1: number analyzed (Participants) | 10
  Month 1 | 5179.0 (930.3)
  Month 3: number analyzed (Participants) | 9
  Month 3 | 4167.8 (642.2)

4. Secondary Outcome: Change From Baseline in ALSFRS-R Total Score at Month 6
Description: ALSFRS-R is a quickly administered (5 minutes) ordinal rating scale that assesses participant's capability and independence in 12 functional activities. All 12 activities, 6 bulbar-respiratory functions, 3 upper extremity functions (writing, cutting food, and dressing), 2 lower-extremity functions (walking and climbing), and 1 other function (turning in bed), are relevant in ALS. Each activity was recorded to the closest approximation from a list of 5 choices, scored 0-4, with the total score ranging from 48 (normal function) to 0 (unable to attempt the task).
Time Frame: Baseline, Month 6
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EPI-589
Number analyzed (Participants) | 14
units on a scale | -4.1 (4.03)

5. Secondary Outcome: Change From Baseline in Vital Capacity at Month 6
Description: Vital capacity is the maximum amount of air a participant can expel from the lungs after a maximum inhalation.
Time Frame: Baseline, Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of capacity
Arm/Group | EPI-589
Number analyzed (Participants) | 14
percentage of capacity | -3.1 (9.36)

6. Secondary Outcome: Change From Baseline in MIP at Month 6
Description: MIP is a measure of the strength of inspiratory muscles, primarily the diaphragm, and allows for the assessment of ventilatory failure, restrictive lung disease, and respiratory muscle strength.
Time Frame: Baseline, Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | EPI-589
Number analyzed (Participants) | 14
cm H2O | 2.4 (24.83)

7. Secondary Outcome: Change From Baseline in Respiratory Rate at Month 6
Description: Respiratory rate is the rate at which breathing occurs.
Time Frame: Baseline, Month 6
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure. 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | EPI-589
Number analyzed (Participants) | 14
breaths/minute
  Sitting | 0.3 (3.45)
  After 5 minutes supine: number analyzed (Participants) | 11
  After 5 minutes supine | -0.6 (5.57)
  After 10 minutes supine: number analyzed (Participants) | 13
  After 10 minutes supine | 0.0 (4.32)

8. Secondary Outcome: Change From Baseline in Heart Rate at Month 6
Description: The heart rate measures the number of times the heart beats per minute.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | EPI-589
Number analyzed (Participants) | 14
beats/minute
  Sitting | 5.2 (10.74)
  After 5 minutes supine: number analyzed (Participants) | 11
  After 5 minutes supine | 7.1 (7.49)
  After 10 minutes supine: number analyzed (Participants) | 13
  After 10 minutes supine | 7.2 (8.39)

9. Secondary Outcome: Change From Baseline in SpO2 at Month 6
Description: SpO2, also known as oxygen saturation, is a measure of the amount of oxygen-carrying hemoglobin in the blood relative to the amount of hemoglobin not carrying oxygen.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | EPI-589
Number analyzed (Participants) | 14
percentage of hemoglobin
  Sitting | -1.0 (1.71)
  After 5 minutes supine: number analyzed (Participants) | 11
  After 5 minutes supine | -0.8 (4.64)
  After 10 minutes supine: number analyzed (Participants) | 13
  After 10 minutes supine | -0.1 (3.55)

10. Secondary Outcome: Change From Baseline in ETCO2 at Month 6
Description: ETCO2 is the amount of CO2 in exhaled air, which assesses ventilation.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of CO2
Arm/Group | EPI-589
Number analyzed (Participants) | 14
percentage of CO2
  Sitting | 2.384 (8.2343)
  After 5 minutes supine: number analyzed (Participants) | 11
  After 5 minutes supine | 0.605 (5.0262)
  After 10 minutes supine: number analyzed (Participants) | 13
  After 10 minutes supine | 7.112 (9.6591)

11. Secondary Outcome: Failure to Thrive: Number of Participants With Weight Loss of More Than 5 Percent (%) From Baseline at Month 6
Description: The failure to thrive as measured by body weight was defined as weight loss of more than 5% from baseline
Time Frame: Baseline, Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | EPI-589
Number analyzed (Participants) | 14
Participants | 2

12. Secondary Outcome: Change From Baseline in Average Solid Swallowing Time and Water Swallowing Time at Month 6
Description: Participants were observed and timed swallowing water as well as solid foods in accordance with a standardized protocol.
Time Frame: Baseline, Month 6
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Number analyzed' signifies participants evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | EPI-589
Number analyzed (Participants) | 19
seconds
  Average Solid Swallowing Time: number analyzed (Participants) | 14
  Average Solid Swallowing Time | 4.80 (11.718)
  Average Water Swallowing Time: number analyzed (Participants) | 13
  Average Water Swallowing Time | 6.65 (20.950)

13. Secondary Outcome: Change From Baseline in Muscle Function at Month 6, as Assessed by Handheld Dynamometry Parameters (Grip Strength, Shoulder Flexion, Knee Extension, Hip Flexion, Elbow Flexion, Elbow Extension, and Ankle Dorsi Flexion)
Description: The strength of designated muscle groups was measured using handheld dynamometry.
Time Frame: Baseline, Month 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | EPI-589
Number analyzed (Participants) | 14
kilograms
  Grip - Left: number analyzed (Participants) | 13
  Grip - Left | -9.69 (15.330)
  Grip - Right: number analyzed (Participants) | 13
  Grip - Right | -7.28 (7.207)
  Shoulder Flexion - Left: number analyzed (Participants) | 12
  Shoulder Flexion - Left | -4.53 (6.922)
  Shoulder Flexion - Right: number analyzed (Participants) | 12
  Shoulder Flexion - Right | -5.43 (8.915)
  Knee Extension - Left | -5.42 (10.254)
  Knee Extension - Right | -5.05 (11.505)
  Knee Flexion - Left | -4.63 (8.237)
  Knee Flexion - Right | -4.01 (9.170)
  Hip Flexion - Left | -6.84 (12.579)
  Hip Flexion - Right | -5.60 (9.627)
  Elbow Flexion - Left: number analyzed (Participants) | 13
  Elbow Flexion - Left | -4.84 (8.377)
  Elbow Flexion - Right: number analyzed (Participants) | 13
  Elbow Flexion - Right | -3.28 (8.186)
  Elbow Extension - Left: number analyzed (Participants) | 13
  Elbow Extension - Left | -5.77 (10.511)
  Elbow Extension - Right: number analyzed (Participants) | 13
  Elbow Extension - Right | -4.28 (9.048)
  Ankle Dorsi Flexion - Left: number analyzed (Participants) | 13
  Ankle Dorsi Flexion - Left | -6.12 (7.609)
  Ankle Dorsi Flexion - Right: number analyzed (Participants) | 13
  Ankle Dorsi Flexion - Right | -4.89 (7.529)

14. Secondary Outcome: Change From Baseline in Number of Words Participant Read at Month 6
Description: The participant performed tasks in which speech was assessed through a perceptual assessment of overall intelligibility, vocal quality, and other factors by a speech language pathologist.
Time Frame: Baseline, Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: words
Arm/Group | EPI-589
Number analyzed (Participants) | 13
words | 0.0 (0.00)

15. Secondary Outcome: Change From Baseline in Time Spent in Reading at Month 6
Description: as for outcome 14
Time Frame: Baseline, Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | EPI-589
Number analyzed (Participants) | 13
seconds | 5.5 (11.78)

16. Secondary Outcome: Change From Baseline in Number of Words Per Minute Read at Month 6
Description: as for outcome 14
Time Frame: Baseline, Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: words/minute
Arm/Group | EPI-589
Number analyzed (Participants) | 13
words/minute | -147.535 (26.7792)

17. Secondary Outcome: Number of Participants With Normal Loudness, Normal Nasality, and Normal Intelligibility
Description: as for outcome 14
Time Frame: Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | EPI-589
Number analyzed (Participants) | 13
Participants
  Normal Loudness | 10
  Normal Nasality | 6
  Normal Intelligibility | 6

18. Secondary Outcome: Level of Disease-Related Biomarker (Glutathione) in Plasma
Description: Glutathione lowest limit of quantification (LLOQ) = 0.089 micromoles (uM) and upper limit of quantification (ULOQ) = 13.916 uM in plasma.
Time Frame: Baseline up to Month 6
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Overall number of participants analyzed' signifies participants with both baseline and Month 6 glutathione in plasma data.
Measure: Mean (Full Range); unit: µM
Arm/Group | EPI-589
Number analyzed (Participants) | 15
µM
  Baseline | 1.34 [0.41 to 2.15]
  Month 6 | 2.73 [0.83 to 11.74]

19. Secondary Outcome: Level of Disease-Related Biomarker (Glutathione) in Cerebrospinal Fluid (CSF)
Description: Glutathione LLOQ = 0.002 uM and ULOQ = 0.35 uM in CSF.
Time Frame: Baseline up to Month 3
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Overall number of participants analyzed' signifies participants with both baseline and Month 3 glutathione in CSF data.
Measure: Mean (Full Range); unit: µM
Arm/Group | EPI-589
Number analyzed (Participants) | 10
µM
  Baseline | 0.13 [0.04 to 0.31]
  Month 3 | 0.13 [0.06 to 0.31]

20. Secondary Outcome: Level of Disease-Related Biomarker (Glutathione) in Urine
Description: Glutathione LLOQ = 0.01 uM, and ULOQ = 1.39 uM in urine.
Time Frame: Baseline up to Month 6
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Overall number of participants analyzed' signifies participants with both baseline and Month 6 glutathione in urine data.
Measure: Mean (Full Range); unit: µM
Arm/Group | EPI-589
Number analyzed (Participants) | 14
µM
  Baseline | 0.12 [0.03 to 0.46]
  Month 6 | 0.17 [0.02 to 0.82]

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) to Month 6
Description: Safety population included any participant who received at least 1 dose of EPI-589.
Arm/Group | EPI-589
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 15/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EPI-589 (N=19)
Aortic valve incompetence (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Eye pain (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Salivary hypersecretion (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 2
Fatigue (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Clostridium difficile infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 5
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aura (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Hypokinesia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT02460679/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02460679/SAP_002.pdf